CLINICAL TRIAL: NCT06967558
Title: The Role of Islet GLP-1 in the Pathogenesis of Prediabetes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adrian Vella, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 24-007677
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: PreDiabetes
Keywords: Impaired Fasting Glucose; Impaired Glucose Tolerance; GLP-1
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance | interventions — exendin (9-39); Sodium Chloride

STUDY DESIGN:
Intervention Model Description: we will study people with normal glucose tolerance with or without impaired fasting glucose together with people with impaired fasting glucose with or without impaired glucose tolerance. All subjects will be studied on 2 occasions - on one they will receive exendin 9-39 and on the other saline
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Exendin 9-39 (Active Comparator): Subjects will receive exendin 9-39 during the study
  Interventions: Biological: Exendin 9-39
- Saline (Placebo Comparator): Subjects will receive saline during the study
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: Exendin 9-39 — Exendin 9-39 is a competitive antagonist of the GLP-1 receptor
  Arms: Exendin 9-39
Biological: Saline — Saline
  Arms: Saline

SUMMARY:
We recently demonstrated that blockade of Glucagon-Like Peptide-1's (GLP-1) receptor (GLP1R) results in changes in islet function without changes in circulating GLP-1. These effects are more pronounced in people with early type 2 diabetes (T2DM) in keeping with increased expression of PC-1/3 and GLP-1 that is observed in diabetic islets. However, its regulation is at present unknown. At present it is unknown if these abnormalities develop in prediabetes and whether they contribute to the phenotypes observed. In this experiment we will use blockade of GLP1R to probe the contribution of endogenous GLP-1 secretion to the regulation of fasting glucose and islet function in prediabetes.

DETAILED DESCRIPTION:
We recently demonstrated that blockade of Glucagon-Like Peptide-1's (GLP-1) receptor (GLP1R) results in changes in islet function without changes in circulating GLP-1. This supports other evidence (rodents and humans) that through the (inducible) expression of a prohormone convertase (PC-1/3), the α-cell can process proglucagon to intact GLP-1. 'Islet' or 'pancreatic' GLP-1 acts in a paracrine fashion to regulate insulin and glucagon secretion. These effects are more pronounced in people with early type 2 diabetes (T2DM). Although pancreatic GLP-1 adapts to support islet function in T2DM, it is unclear if this mechanism is upregulated in prediabetes and whether it contributes to the phenotype(s) observed. Abnormal α-cell responsivity to glucose, measured using G50, is associated with Impaired Fasting Glucose (IFG); β-cell dysfunction is associated with Impaired Glucose Tolerance (IGT). Does IGT (or IFG) represent selective failure of intra-islet GLP-1 to support islet function? In this experiment we will use blockade of GLP1R to probe the contribution of endogenous GLP-1 secretion to the regulation of fasting glucose and islet function in prediabetes

ELIGIBILITY:
Inclusion Criteria:

* People with stable weight and no history of diabetes.
* Fasting glucose < 126 mg/dL
* 2hr glucose after 75g OGTT < 200 mg/dL

Exclusion Criteria:

* Age < 25 or > 70 years (to avoid studying subjects who could have latent type 1 diabetes, or the effects of age extremes in subjects with normal or impaired fasting glucose).
* HbA1c > 6.5%
* Use of any glucose-lowering agents including metformin or sulfonylureas.
* For female subjects: positive pregnancy test at the time of enrollment or study
* History of prior upper abdominal surgery such as adjustable gastric banding, pyloroplasty and vagotomy.
* Active systemic illness or malignancy.
* Symptomatic macrovascular or microvascular disease.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Alpha-cell responsivity to glucose as measured by G50 | 0-240 minutes
  The change in glucose necessary to suppress glucagon secretion by 50%
Beta-cell responsivity to glucose | 0-240 minutes
  This is measured as the gradient of the increase in insulin secretion rate per unit increase in glucose concentration

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No